CLINICAL TRIAL: NCT01937715
Title: An Open-Label, Multi-Center, Randomized Phase 1b/2 Study Of PF-05212384 Plus 5-Fluorouracil-Leucovorin-Irinotecan (FOLFIRI) Versus Bevacizumab Plus FOLFIRI In Metastatic Colorectal Cancer
Brief Title: A Study Of PF-05212384 Plus FOLFIRI Versus Bevacizumab Plus FOLFIRI In Metastatic Colorectal Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: B2151007 was prematurely discontinued due to Pfizer's change in prioritization for the portfolio and is not due to any safety concerns or regulatory interaction
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2151007; 2013-002096-18 (EudraCT Number)
Record Dates: First submitted 2013-08-27; First posted 2013-09-09 (Estimated); Results first posted 2016-08-18 (Estimated); Last update posted 2016-08-18 (Estimated); Status verified 2016-07

CONDITIONS: Metastatic Colorectal Carcinoma
MeSH Terms: conditions — Colorectal Neoplasms | interventions — gedatolisib; Bevacizumab; IFL protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Experimental): PF-05212384 plus FOLFIRI
  Interventions: Drug: PF-05212384; Drug: FOLFIRI regimen
- Arm B (Active Comparator): Bevacizumab plus FOLFIRI
  Interventions: Biological: Bevacizumab; Drug: FOLFIRI

INTERVENTIONS:
Drug: PF-05212384 — PF-05212384 at the Recommended phase 2 dose (RP2D/MTD) weekly
  Arms: Arm A
Drug: FOLFIRI regimen — The RP2D/MTD dose of FOLFIRI regimen every 2 weeks
  Arms: Arm A
Biological: Bevacizumab — 5 mg/m^2 every 2 weeks or 7.5 mg/m^2 every 3 weeks
  Arms: Arm B
Drug: FOLFIRI — Full dose FOLFIRI regimen every 2 weeks
  Arms: Arm B

SUMMARY:
This is a multicenter, open label Phase 1b/2 study in patients with metastatic colorectal carcinoma. The Phase 1b will identify the dose of the combination of PF-05212384 plus FOLFIRI. The randomized, two-arm Phase 2 portion will compare the efficacy and safety of PF-05212384 plus FOLFIRI to that of bevacizumab plus FOLFIRI.

The study population will consist of patients with mCRC previously treated with an oxaliplatin-based regimen in the first line setting or who have progressed within 6 months of the end of an adjuvant oxaliplatin-based regimen.

ELIGIBILITY:
Inclusion Criteria:

* Advanced colorectal carcinoma.
* Progression on prior oxaliplatin-containing regimen used in 1st line setting for mCRC or progression within 6 months of end of oxaliplatin-containing regimen in the adjuvant setting.
* Tumor tissue available at time of screening for molecular profiling.
* Adequate performance status.
* Adequate glucose control, bone marrow, kidney, liver, and heart function.

Exclusion Criteria:

* Participation in other studies involving investigational drug(s) (Phases 1-4) before the current study begins and/or during study participation.
* Prior irinotecan treatment.
* Prior radiation to the pelvis or abdomen in the metastatic or locally advanced setting.
* History of Gilbert's syndrome.
* Active brain metastases.
* Deep vein thrombosis in the preceding 2 months.
* History of interstitial lung disease.
* RAS (KRAS/NRAS) wild type mCRC not previously treated with an anti-EGFR containing regimen (unless contraindicated or not considered standard practice per clinical site or country guidelines).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-02; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (38):
- United States (34):
  - St. Jude Hospital Yorba Linda DBA St. Joseph Heritage Healthcare, Fullerton, California
  - UCLA Hematology Oncology, Irvine, California
  - Drug Management Only: UCLA West Medical Pharmacy, Attn Steven L. Wong, Pharm .D., Los Angeles, California
  - Drug Management Only: UCLA West Medical Pharmacy, Los Angeles, California
  - UCLA West Medical Pharmacy, Att: Steven L. Wong, Pharm D., Los Angeles, California
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - Ronald Regan UCLA Medical Center, Drug Information Center, Los Angeles, California
  - TRIO-US Central Administration, Regulatory Management Only, Los Angeles, California
  - TRIO-US Central Administration, Los Angeles, California
  - TRIO_US, Los Angeles, California
  - UCLA Hematology Oncology Administrative Address, Los Angeles, California
  - Westwood Bowyer Clinic, Peter Morton Medical Building, Los Angeles, California
  - West Valley Hematology/Oncology Med Group, Northridge, California
  - UCLA/Pasadena Healthcare, Pasadena, California
  - Central Coast Medical Oncology Corporation, Santa Maria, California
  - UCLA Hematology Oncology, Santa Monica, California
  - UCLA Santa Monica Medical Center & Orthopaedic Hospital, Santa Monica, California
  - UCLA/Santa Clarita Valley Cancer Center, Valencia, California
  - UCLA Cancer Center, Westlake Village, California
  - Comprehensive Cancer Centers of Nevada Research Department, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada, Henderson, Nevada
  - Comprehensive Cancer Centers of NV, Las Vegas, Nevada
  - COmprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Comprehensive Cancer Centers for Nevada, Las Vegas, Nevada
  - Metrohealth Medical Center, Cleveland, Ohio
  - Medical Group of the Carolinas - Hematology Spartanburg, Spartanburg, South Carolina
  - Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Kadlec Medical Center, Richland, Washington
  - Outpatient Imaging Center, Richland, Washington
  - Investigational Drug Services, Seattle, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Medical Oncology Associates, PS, Spokane, Washington
  - Spokane Valley Cancer Center, Spokane Valley, Washington
- Canada (2):
  - The Ottawa Hospital Cancer Centre, Ottawa, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
- Spain (2):
  - Hospital Universitari Vall d'Hebron, Barcelona, Spain
  - Hospital General Universitario Gregorio Marañón, Madrid, Spain

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B2151007&StudyName=A%20Study%20Of%20PF-05212384%20Plus%20FOLFIRI%20Versus%20Bevacizumab%20Plus%20FOLFIRI%20In%20Metastatic%20Colorectal%20Cancer%20

RESULTS

PARTICIPANT FLOW:
Groups:
- PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 1: Participants received intravenous (IV) infusion of PF-05212384 90 mg weekly and IV infusions of irinotecan 150 mg/m^2, leucovorin 320 mg/m^2, 5- fluorouracil (FU) 1920 mg/m^2, and IV bolus of 5-FU 320 mg/m^2 on Days 1 and 15 of each cycle.
- PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 2A: Participants received intravenous (IV) infusion of PF-05212384 90 mg weekly and IV infusions of irinotecan 180 mg/m^2, leucovorin 400 mg/m^2, 5- fluorouracil (FU) 2400 mg/m^2, and IV bolus of 5-FU 400 mg/m^2 on Days 1 and 15 of each cycle.
- PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 2B: Participants received intravenous (IV) infusion of PF-05212384 110 mg weekly and IV infusions of irinotecan 180 mg/m^2, leucovorin 400 mg/m^2, 5- fluorouracil (FU) 2400 mg/m^2, and IV bolus of 5-FU 400 mg/m^2 on Days 1 and 15 of each cycle.
- PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 3: Participants received intravenous (IV) infusion of PF-05212384 130 mg weekly and IV infusions of irinotecan 180 mg/m^2, leucovorin 400 mg/m^2, 5- fluorouracil (FU) 2400 mg/m^2, and IV bolus of 5-FU 400 mg/m^2 on Days 1 and 15 of each cycle.
- PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 4: Participants received intravenous (IV) infusion of PF-05212384 150 mg weekly and IV infusions of irinotecan 180 mg/m^2, leucovorin 400 mg/m^2, 5- fluorouracil (FU) 2400 mg/m^2, and IV bolus of 5-FU 400 mg/m^2 on Days 1 and 15 of each cycle.
Period: Overall Study
Arm/Group | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 1 | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 2A | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 2B | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 3 | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 4
Started | 3 | 4 | 3 | 5 | 3
Completed | 3 | 3 | 3 | 1 | 1
Not Completed | 0 | 1 | 0 | 4 | 2
Not completed — Death | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 2
Not completed — Other | 0 | 0 | 0 | 3 | 0

BASELINE CHARACTERISTICS:
Population: The baseline analysis population included all participants who received at least 1 dose of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 1 | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 2A | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 2B | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 3 | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 4 | Total
Number analyzed (Participants) | 3 | 4 | 3 | 5 | 3 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.7 (11.7) | 54.3 (10.1) | 63.3 (11.6) | 65.8 (9) | 54.3 (5.5) | 56.9 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 0 | 0 | 3 | 7
  Male | 2 | 1 | 3 | 5 | 0 | 11

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Dose-Limiting Toxicities (DLTs) in First Cycle of Therapy
Description: DLTs were classified according to Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 and defined as any of the following events judged to be attributed to the combination of PF-05212384 plus FOLFIRI: hematologic (febrile neutropenia or a sustained temperature >=38 degrees Celcius for >1 hour, grade >=3 neutropenic infection, grade 3 thrombocytopenia with bleeding, grade 4 thrombocytopenia); non-hematologic (grade >=2 pneumonitis, grade >=3 toxicities, toxicities which resulted in failure to deliver at least 75% of the planned total dose of PF-05212384 and/or 50% of the planned total dose of FOLFIRI during the first cycle, toxicities which resulted in delay of start of Cycle 2 by >2 weeks of scheduled day (Day 43 of study), Grade 3 QTc prolongation).
Time Frame: Day 1 up to Day 28
Population: The dose limiting toxicity analysis set included participants in Phase 1B who started treatment and who did not have a major treatment deviation in the lead-in period and the first cycle of treatment.
Measure: Number; unit: percentage of participants
Arm/Group | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 1 | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 2A | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 2B | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 3 | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 4
Number analyzed (Participants) | 3 | 4 | 3 | 5 | 3
percentage of participants | 0 | 0 | 0 | 20.0 | 66.7

2. Primary Outcome: Progression-Free Survival (PFS)
Description: Progression-free survival was the time from randomization the date to date of first documentation of progression or death due to any cause, whichever occurred first. Documentation of progression was by objective disease assessment as defined by the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
Time Frame: Baseline (Day 1) up to disease progression or death whichever occurred first (up to 18 months)
Population: PFS was the primary efficacy endpoint for the study and was only to be assessed in the Phase 2 portion of the study. As this study was terminated due to Pfizer portfolio prioritization prior to the Phase 2 portion, there are no efficacy evaluations for Phase 2.
Arm/Group | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 1 | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 2A | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 2B | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 3 | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 4
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Number of Participants With Best Overall Response (Phase 1B)
Description: Best overall response is defined as the best response recorded from randomization (or first dose for patients in the Phase 1B) until disease progression, death, start of new anti-cancer treatment or end of study. The categories for best overall response include: complete response (CR) (complete disappearance of all target lesions with the exception of nodal disease and all target nodes must decrease to normal size (short axis <10 millimeters (mm)); partial response (PR) (at least a 30 percent (%) decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters); stable disease (SD) (not qualify for CR, PR or Progression); progressive disease (PD) (20% increase in the sum of diameters of target measurable lesions above the smallest sum observed (over baseline if no decrease in the sum is observed during therapy), with a minimum absolute increase of 5 mm); indeterminate (IND) (progression has not been documented).
Time Frame: Every 8 weeks from Cycle 1 Day 1 until 28 days of last dose
Population: All participants in the full analysis (FA) set who had measureable disease and an adequate baseline assessment of the disease.
Measure: Number; unit: participants
Arm/Group | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 1 | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 2A | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 2B | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 3 | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 4
Number analyzed (Participants) | 2 | 4 | 3 | 5 | 3
participants
  PD | 2 | 2 | 0 | 1 | 1
  SD | 0 | 2 | 2 | 3 | 0
  PR | 0 | 0 | 1 | 0 | 0
  Indeterminant | 0 | 0 | 0 | 1 | 2

4. Secondary Outcome: Number of Participants With All Causality Treatment-Emergent Adverse Events (AEs), Serious Adverse Events (SAEs), and Discontinuations by Relationship and Seriousness
Description: An AE was any untoward medical occurrence without regard to causality in a participant who received study drug. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. An AE was considered treatment emergent if the event occurred for the first time after the start of study treatment and within 28 days after final dose of study treatment and was not seen prior to the start of treatment; or the event was seen prior to the start of treatment but increased in CTCAE version 4.0 grade after the start of study treatment and within 28 days after final dose of study treatment.
Time Frame: Baseline up to final study evaluation (within 28 days of last dose)
Population: All participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 1 | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 2A | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 2B | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 3 | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 4
Number analyzed (Participants) | 3 | 4 | 3 | 5 | 3
participants
  Number (#) of Participants with AEs | 3 | 4 | 3 | 5 | 3
  # of Participants with SAEs | 0 | 0 | 2 | 2 | 3
  # of Participants with Grade 3 or 4 AEs | 0 | 3 | 3 | 3 | 3
  # of Participants with Grade 5 AEs | 0 | 0 | 0 | 0 | 0
  # of Participants D/C'd Study Due to AEs | 0 | 0 | 0 | 0 | 0
  # of Participants D/C'd PF-05212384 Due to AEs | 0 | 0 | 0 | 0 | 1
  Number of Participants D/C'd FOLFIRI Due to AEs | 0 | 0 | 0 | 0 | 1

5. Secondary Outcome: Number of Participants With All Causality AEs by System Organ Class (SOC)
Description: An AE was any untoward medical occurrence without regard to causality in a participant who received study drug.
Time Frame: Baseline up to final study evaluation (within 28 days of last dose)
Population: All participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 1 | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 2A | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 2B | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 3 | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 4
Number analyzed (Participants) | 3 | 4 | 3 | 5 | 3
participants
  Blood and lymphatic system disorders | 0 | 2 | 0 | 1 | 0
  Eye disorders | 0 | 1 | 0 | 0 | 1
  Gastrointestinal disorders | 3 | 4 | 3 | 5 | 3
  General disorders & administration site conditions | 2 | 2 | 2 | 4 | 2
  Hepatobiliary disorders | 0 | 0 | 0 | 1 | 0
  Immune system disorders | 0 | 0 | 1 | 0 | 0
  Infections and infestations | 1 | 3 | 1 | 1 | 1
  Injury, poisoning and procedural complications | 0 | 3 | 0 | 0 | 0
  Investigations | 1 | 4 | 1 | 2 | 2
  Metabolism and nutrition disorders | 2 | 3 | 1 | 3 | 2
  Musculoskeletal and connective tissue disorders | 1 | 4 | 1 | 1 | 1
  Nervous system disorders | 0 | 2 | 3 | 2 | 1
  Psychiatric disorders | 3 | 2 | 0 | 0 | 2
  Renal and urinary disorders | 0 | 2 | 0 | 1 | 0
  Respiratory, thoracic and mediastinal disorders | 1 | 1 | 3 | 3 | 1
  Skin and subcutaneous tissue disorders | 1 | 3 | 2 | 2 | 3
  Vascular disorders | 0 | 1 | 1 | 1 | 1

6. Secondary Outcome: Number of Participants With Treatment-Emergent AEs by Worst On-Study Grade
Description: An AE was any untoward medical occurrence without regard to causality in a participant who received study drug. AE grades were defined according to Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 criteria.
Time Frame: Baseline up to final study evaluation (within 28 days of last dose)
Population: All participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 1 | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 2A | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 2B | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 3 | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 4
Number analyzed (Participants) | 3 | 4 | 3 | 5 | 3
participants
  Any AEs, Grade 1 | 0 | 0 | 0 | 1 | 0
  Any AEs, Grade 2 | 3 | 1 | 0 | 1 | 0
  Any AEs, Grade 3 | 0 | 3 | 3 | 2 | 3
  Any AEs, Grade 4 | 0 | 0 | 0 | 1 | 0
  Any AEs, Grade 5 | 0 | 0 | 0 | 0 | 0
  Any AEs, total | 3 | 4 | 3 | 5 | 3

7. Secondary Outcome: Number of Participants With Hematological Test Abnormalities
Description: Number of participants with NCI CTCAE version 4.0 grade 1 to 4 hematological test abnormalities.
Time Frame: Day 1 and Day 15 of each cycle
Population: All participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 1 | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 2A | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 2B | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 3 | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 4
Number analyzed (Participants) | 3 | 4 | 3 | 5 | 2
participants
  Anemia | 3 | 4 | 3 | 5 | 2
  Hemoglobin increased | 0 | 0 | 0 | 0 | 0
  Lymphocyte count increased | 0 | 1 | 0 | 0 | 0
  Lymphopenia | 2 | 2 | 2 | 3 | 0
  Neutrophils (Absolute) | 0 | 4 | 2 | 2 | 2
  Platelets | 0 | 2 | 0 | 2 | 0
  White blood cells | 1 | 3 | 3 | 3 | 2

8. Secondary Outcome: Number of Participants With Coagulation Test Abnormalities
Description: Number of participants with NCI CTCAE version 4.0 grade 1 to 4 Coagulation test abnormalities.
Time Frame: Day 1 and Day 15 of Cycle 1, Day 1 of Cycle 2 and subsequent cycles
Population: All participants who received at least 1 dose of study medication. n=number of participants evaluated against criteria.
Measure: Number; unit: participants
Arm/Group | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 1 | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 2A | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 2B | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 3 | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 4
Number analyzed (Participants) | 3 | 4 | 3 | 5 | 3
participants
  Partial thromboplastin time (N=3, 4, 3, 5, 2) | 1 | 0 | 1 | 2 | 2
  Prothrombin time (PT) (N=3, 3,2, 5, 1) | 1 | 0 | 2 | 1 | 1
  PT INR (N=3, 4, 3, 5, 2) | 1 | 0 | 2 | 0 | 1

9. Secondary Outcome: Number of Participants With Chemistry Test Abnormalities
Description: Number of participants with NCI CTCAE version 4.0 grade 1 to 4 Chemistry test abnormalities.
Time Frame: Day 1 and Day 15 of each cycle
Population: All participants who received at least 1 dose of study medication. n=number of participants evaluated against criteria.
Measure: Number; unit: participants
Arm/Group | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 1 | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 2A | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 2B | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 3 | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 4
Number analyzed (Participants) | 3 | 4 | 3 | 5 | 2
participants
  Alanine aminotransferase | 0 | 1 | 1 | 3 | 1
  Alkaline phosphatase | 3 | 2 | 0 | 3 | 1
  Aspartate aminotransferase | 2 | 2 | 2 | 4 | 1
  Bilirubin (total) | 0 | 2 | 0 | 1 | 0
  Creatinine | 1 | 2 | 3 | 4 | 2
  Hyperglycemia | 2 | 3 | 1 | 5 | 2
  Hypermagnesemia | 0 | 0 | 1 | 0 | 0
  Hypoalbuminemia | 2 | 2 | 0 | 3 | 1
  Hypocalcemia | 0 | 0 | 0 | 2 | 0
  Hypoglycemia | 1 | 0 | 0 | 0 | 0
  Hypokalemia | 2 | 2 | 1 | 0 | 1
  Hypomagnesemia | 0 | 1 | 1 | 1 | 0
  Hyponatremia | 3 | 2 | 1 | 4 | 0
  Hypohphosphatemia | 1 | 0 | 0 | 1 | 0
  Hyperkalemia | 0 | 1 | 0 | 0 | 0

10. Secondary Outcome: Number of Participants With Urinalysis Test Abnormalities
Description: Number of participants with NCI CTCAE version 4.0 grade 1 to 4 Urinalysis test abnormalities.
Time Frame: Day 1 and Day 15 of Cycle 1, Day 1 of Cycle 2 and subsequent cycles
Population: All participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 1 | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 2A | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 2B | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 3 | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 4
Number analyzed (Participants) | 3 | 4 | 3 | 5 | 2
participants | 2 | 1 | 1 | 2 | 2

11. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax): PF-05212384, Irinotecan, and Fluorouracil
Description: Maximum Plasma Concentration of PF-05212384, Irinotecan, and Fluorouracil
Time Frame: PF-05212384: Cycle 1 Day 3. Irinotecan: Cycle 1 Day 1. Fluorouracil: Cycle 1 Day 1.
Population: Randomized participants (or enrolled participants for Phase 1B) who started treatment and who had at least one of the pharmacokinetic parameters of interest estimated.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram (ng)/milliliter (mL)
Arm/Group | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 1 | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 2A | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 2B | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 3 | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 4
Number analyzed (Participants) | 3 | 4 | 3 | 5 | 3
nanogram (ng)/milliliter (mL)
  PF-05212384 (n=3,4,2,5,3) | 8245 (25) | 6554 (66) | 33470 (NA) — Summary statistics were not presented if fewer than 3 subjects had reportable parameter values. Mean value is provided for Dose level 2B. | 8222 (35) | 10250 (11)
  Irinotecan (n=3,4,1,5,3) | 1782 (4) | 1323 (43) | 1550 (NA) — Summary statistics were not presented if fewer than 3 subjects had reportable parameter values. Individual value is provided for Dose level 2B. | 1585 (17) | 1755 (6)
  Fluorouracil (n=3,4,1,4,3) | 18390 (85) | 18950 (41) | 44000 (NA) — Summary statistics were not presented if fewer than 3 subjects had reportable parameter values. Individual value is provided for Dose level 2B. | 26790 (18) | 26920 (3)

12. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax): PF-05212384, Irinotecan, and Fluorouracil
Description: Time to Reach Maximum Observed Plasma Concentration of PF-05212384, Irinotecan, and Fluorouracil
Time Frame: PF-05212384: Cycle 1 Day 3. Irinotecan: Cycle 1 Day 1. Fluorouracil: Cycle 1 Day 1.
Population: as for outcome 11
Measure: Median (Full Range); unit: hour (hr)
Arm/Group | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 1 | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 2A | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 2B | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 3 | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 4
Number analyzed (Participants) | 3 | 4 | 3 | 5 | 3
hour (hr)
  PF-05212384 (n=3,4,2,5,3) | 0.500 [0.450 to 0.500] | 0.550 [0.450 to 0.617] | 0.500 [0.500 to 0.500] | 0.500 [0.383 to 0.500] | 0.500 [0.483 to 1.03]
  Irinotecan (n=3,4,1,5,3) | 2.02 [1.98 to 2.02] | 2.04 [2.00 to 2.15] | 1.95 [1.95 to 1.95] | 2.25 [1.98 to 2.50] | 2.00 [1.98 to 2.02]
  Fluorouracil (n=3,4,1,4,3) | 0.0830 [0.0330 to 0.150] | 0.167 [0.167 to 0.233] | 0.0830 [0.0830 to 0.0830] | 0.125 [0.0670 to 0.250] | 0.150 [0.150 to 46.2]

13. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast): PF-05212384 and Irinotecan
Description: Area Under the Curve From Time Zero to Last Quantifiable Concentration of PF-05212384, and Irinotecan
Time Frame: PF-05212384: Cycle 1 Day 3. Irinotecan: Cycle 1 Day 1.
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 1 | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 2A | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 2B | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 3 | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 4
Number analyzed (Participants) | 3 | 4 | 3 | 5 | 3
ng*hr/mL
  PF-05212384 (n=3,4,1,5,3) | 11460 (22) | 9129 (33) | 30700 (NA) — Summary statistics were not presented if fewer than 3 subjects had reportable parameter values. Individual value is provided for Dose level 2B. | 13570 (40) | 14760 (34)
  Irinotecan (n=3,4,1,4,3) | 12510 (8) | 9164 (53) | 8050 (NA) — Summary statistics were not presented if fewer than 3 subjects had reportable parameter values. Individual value is provided for Dose level 2B. | 10340 (15) | 11030 (28)

14. Secondary Outcome: Area Under the Plasma Concentration-Time Profile From Time 0 Extrapolated to Infinite Time (AUCinf): PF-05212384 and Irinotecan
Description: Area Under the Plasma Concentration-Time Profile From Time 0 Extrapolated to Infinite Time of PF-05212384 and Irinotecan
Time Frame: PF-05212384: Cycle 1 Day 3. Irinotecan: Cycle 1 Day 1.
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 1 | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 2A | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 2B | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 3 | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 4
Number analyzed (Participants) | 3 | 4 | 1 | 5 | 3
ng*hr/mL
  PF-05212384 | 11820 (22) | 9289 (32) | 30900 (NA) — Summary statistics were not presented if fewer than 3 subjects had reportable parameter values. Individual value is provided for Dose level 2B. | 13830 (40) | 15270 (34)
  Irinotecan | 13120 (10) | 9709 (54) | 8350 (NA) — Summary statistics were not presented if fewer than 3 subjects had reportable parameter values. Individual value is provided for Dose level 2B. | 10900 (16) | 11560 (29)

15. Secondary Outcome: Terminal Elimination Half-Life (t1/2): PF-05212384 and Irinotecan
Description: Terminal Elimination Half-Life of PF-05212384 and Irinotecan
Time Frame: PF-05212384: Cycle 1 Day 3. Irinotecan: Cycle 1 Day 1.
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 1 | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 2A | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 2B | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 3 | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 4
Number analyzed (Participants) | 3 | 4 | 1 | 5 | 3
hour
  PF-05212384 | 33.63 (1.3503) | 27.90 (3.3695) | 29.2 (NA) — Summary statistics were not presented if fewer than 3 subjects had reportable parameter values. Individual value is provided for Dose level 2B. | 29.18 (6.9909) | 36.97 (1.9035)
  Irinotecan | 5.127 (0.70692) | 5.533 (1.1621) | 4.97 (NA) — Summary statistics were not presented if fewer than 3 subjects had reportable parameter values. Individual value is provided for Dose level 2B. | 5.360 (0.40817) | 5.107 (0.40427)

16. Secondary Outcome: Number of Participants Meeting Maximum Post-Baseline QTc Interval Values
Description: Criteria for corrected QT interval using Fridericia's formula (QTcF) meeting potential clinical concern included: an absolute value >=450 - <480 msec, >=480-<500 msec, >500 msec; an absolute change 30 - <60, >=60 msec.
Time Frame: Baseline, Cycle 1 Day 1, and Cycle 2 Day 2
Population: All participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 1 | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 2A | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 2B | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 3 | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 4
Number analyzed (Participants) | 3 | 4 | 3 | 5 | 3
participants
  QTcF Interval <450 msec | 3 | 4 | 3 | 3 | 3
  QTcF Interval 450-480 msec | 0 | 0 | 0 | 2 | 0
  QTcF Interval >480-500 msec | 0 | 0 | 0 | 0 | 0
  QTcF Interval >500 msec | 0 | 0 | 0 | 0 | 0
  QTcF Interval increase =< 30 msec | 2 | 3 | 3 | 4 | 3
  QTcF Interval increase >30 to =<60 msec | 1 | 1 | 0 | 1 | 0
  QTcF Interval increase >60 | 0 | 0 | 0 | 0 | 0

17. Secondary Outcome: Number of Participants With Expression of Gene Sequences or Gene Amplications in Biopsied Tumor Tissue
Description: Biomarker evaluation were to be performed on fresh biopsies, as well as on archival biopsies collected during the study. Samples were to be analyzed for biomarkers indicative of pathway modulation or for genetic markers correlated to drug sensitivity.
Time Frame: Baseline and Cycle 2 Day 17
Population: Paired fresh tumor biopsies were only done in 1 subject but not summarized.
Arm/Group | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 1 | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 2A | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 2B | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 3 | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 4
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

18. Secondary Outcome: Number of Participants With Gene and/or Protein Expression Biomarkers Relating to the PI3K and/or mTOR Pathway Activation in Biopsied Tumor Tissue
Description: as for outcome 17
Time Frame: Baseline and Cycle 2 Day 17
Population: Paired fresh tumor biopsies were only done in 1 subject but not summarized.
Arm/Group | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 1 | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 2A | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 2B | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 3 | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 4
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

19. Secondary Outcome: Number of Participants With Best Overall Response (Phase 2)
Description: as for outcome 3
Time Frame: Day 1 up to Day 28
Population: As this study was terminated due to Pfizer portfolio prioritization prior to the Phase 2 portion, there are no efficacy evaluations for Phase 2. No data were collected for Phase 2.
Arm/Group | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 1 | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 2A | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 2B | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 3 | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 4
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

20. Secondary Outcome: Duration of Response (Phase 2)
Description: Duration of response is the time from first documentation of CR or PR to date of first documentation of objective progression or death.
Time Frame: Day 1 to Day 28
Population: as for outcome 19
Arm/Group | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 1 | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 2A | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 2B | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 3 | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 4
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

21. Secondary Outcome: Overall Survival (Phase 2)
Description: Overall survival is the time from randomization date to date of death due to any cause.
Time Frame: Day 1 up to Day 28
Population: as for outcome 19
Arm/Group | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 1 | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 2A | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 2B | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 3 | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 4
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

22. Secondary Outcome: Number of Participants With Evidence of Pathway Signaling Related Genes and/or Proteins in Biopsied Tumor Tissue (Phase 2)
Description: Biomarker evaluation were to be performed on these fresh biopsies, as well as on archival biopsies collected during the study. Samples were to be analyzed for biomarkers indicative of pathway modulation or for genetic markers correlated to drug sensitivity.
Time Frame: Baseline and Cycle 2 Day 17
Population: Levels of signaling proteins in biopsied tumor tissue was the secondary endpoint for the Phase 2 portion of the study. As this study was terminated due to Pfizer portfolio prioritization prior to the Phase 2 portion, no data were collected for Phase 2.
Arm/Group | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 1 | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 2A | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 2B | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 3 | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 4
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

23. Secondary Outcome: Change From Baseline in Functional Assessment of Cancer Therapy-Colorectal (FACT-C) (Phase 2)
Description: The FACT-C was to assess health-related quality of life and colorectal cancer (CRC)-related symptoms. It includes a total of 36 items, which are summarized into 6 subscales: physical well-being (7 items), functional well-being (7 items), social/family well-being (7 items), emotional well-being (6 items), CRC subscale (9 items) which addresses a subset of CRC concerns such as diarrhea.
Time Frame: Day 1 of each cycle
Population: FACT-C was only applicable to the Phase 2 portion of the study. As this study was terminated due to Pfizer portfolio prioritization prior to the Phase 2 portion, no data were collected for Phase 2.
Arm/Group | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 1 | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 2A | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 2B | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 3 | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 4
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline to end of treatment
Arm/Group | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 1 | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 2A | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 2B | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 3 | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 4
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/4 | 2/3 | 2/5 | 3/3
Other Adverse Events (participants affected / at risk) | 3/3 | 4/4 | 3/3 | 5/5 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 1 (N=3) | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 2A (N=4) | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 2B (N=3) | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 3 (N=5) | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 4 (N=3)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Anal fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Periorbital infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 1 (N=3) | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 2A (N=4) | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 2B (N=3) | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 3 (N=5) | PF-05212384+5-FU+Irinotecan+Leucovorin:Dose Level 4 (N=3)
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0 | 0
Eye disorder (Eye disorders) | 0 | 0 | 0 | 0 | 1
Vision blurred (Eye disorders) | 0 | 1 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 2 | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 3 | 3 | 3 | 3
Dry mouth (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Lip disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Lip swelling (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 2 | 1 | 3 | 3
Oral dysaesthesia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Paraesthesia oral (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Proctalgia (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 2 | 1 | 3 | 2
Tongue coated (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 2 | 0 | 2 | 2
Asthenia (General disorders) | 0 | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 0 | 0
Chills (General disorders) | 0 | 1 | 0 | 0 | 0
Early satiety (General disorders) | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 1 | 2 | 2 | 2 | 1
Mucosal inflammation (General disorders) | 1 | 0 | 1 | 1 | 1
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 1 | 0 | 1 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0 | 0
Candida infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Periorbital infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 1
Blood albumin decreased (Investigations) | 0 | 1 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 1 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 4 | 1 | 0 | 2
Platelet count decreased (Investigations) | 0 | 2 | 0 | 0 | 0
Weight decreased (Investigations) | 1 | 0 | 0 | 2 | 1
White blood cell count decreased (Investigations) | 0 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 3 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Disturbance in attention (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Head discomfort (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 2 | 1 | 1 | 1
Lethargy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Derailment (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 2 | 2 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 1 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 1 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Flushing (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
As this study was terminated due to Pfizer portfolio prioritization prior to the Phase 2 portion, there are no efficacy evaluations for Phase 2.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.